CLINICAL TRIAL: NCT00353639
Title: Telomere Repair Gene Mutations in Inflammatory Bowel Disease
Brief Title: Telomere Repair Gene Mutation in Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060082; 06-H-0082
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Disease
Keywords: Ulcera; Telomerase; TERT; TERC; SBDS; DNA Helicase; Inflammatory Bowel Disease; IBD
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- IBD subjects: Subjects with Inflammatory Bowell Disease

SUMMARY:
This study will evaluate and compare the genes of the telomere repair complex in healthy control subjects, patients with blood diseases, and patients with inflammatory bowel disease to identify what, if any, changes are associated specifically with inflammatory bowel disease.

Patients between 2 and 80 years of age with ulcerative colitis or regional enteritis may be eligible for this study. Participants are recruited from the practice of Dr. Stuart Danovitch, Washington, D.C.

Researchers have established that minor differences in a specific set of genes called the telomere repair complex are related to immune-mediated diseases of the bone marrow. NIH researchers are now interested in whether inflammatory bowel disease and other autoimmune diseases show a similar pattern of genetic differences.

Participants provide a cell sample for evaluation of the telomere repair complex. The sample is collected via buccal swab, a gentle scraping of the inside of the cheek, and stored for use in research.

DETAILED DESCRIPTION:
We have identified inherited mutations in genes of the telomere repair complex in patients with acquired aplastic anemia. These mutations diminish the ability of cells to repair the ends of chromosomes, called telomeres, which normally shorten with each cell division. Mutations in TERC, the gene which encodes for the RNA template of the complex; in TERT, the gene for the enzyme in the complex, and also in the Schwachman-Bodian-Diamond syndrome gene (SBDS), which we believe to be associated with telomere repair, lead to reduced telomerase activity, diminished numbers of hematopoietic cells in the bone marrow, and presumably also a deficiency in the ability of cells to respond to immunological attack and destruction of the hematopoietic system.

This laboratory research protocol will allow us to evaluate whether similar gene mutations might underlie other autoimmune diseases, here specifically, inflammatory bowel disease, which share broad pathophysiologic features with immune-mediated aplastic anemia. We will directly assess by DNA sequencing suspect genes (TERC, TERT, SBDS, DNA helicases and others) in buccal mucosal samples obtained from patients with inflammatory bowel disease (IBD). Analyses from large numbers of controls have defined polymorphisms for these genes. IBD samples will allow us to determine whether mutations in these genes are more prevalent in this patient population and to test the hypotheses that telomere repair defects underlie human autoimmunity, or that these genes are specifically involved in hematology as risks factors for bone marrow failure.

ELIGIBILITY:
* INCLUSION CRITERIA:

Diagnosis of ulcerative colitis or regional enteritis

For adults:

Ability to comprehend the investigational nature of the study and provide informed consent. Or

For minors: Written informed consent from one parent or guardian and informed assent. The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

Age greater than 2 but less or equal to 80 years old

EXCLUSION CRITERIA:

All subjects not fulfilling the inclusion criteria will be considered ineligible.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with Inflammatory Bowell Disease
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2006-05-15 (Actual); Primary Completion 2006-05-15 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
To identify if telomere repair complex gene mutations are abnormally prevalent among patients with IBO. | Ongoing
  To identify if telomere repair complex gene mutations are abnormally prevalent among patients with IBO.

SECONDARY OUTCOMES:
To correlate telomere repair gene mutations in subjects with immune mediated disease stratified based on diagnosis as they relate to clinical course and response to therapy. | Ongoing
  We aim to correlate telomere repair gene mutations in subjects with immune mediated disease stratified based on diagnosis with clinical course and response to therapy.
To compare the telomere repair gene mutations of normal individuals (from large populations studies in the public domain) as well as to those of patients with known bone marrow failure | Ongoing
  We aim to compare the telomere repair gene mutations of normal individuals with those of patients with known bone marrow failure

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-H-0082.html